CLINICAL TRIAL: NCT03576079
Title: Effect of Laser Irradiation Versus Anterior Repositioning Splint in Treatment of Disc Displacement With Reduction A Randomized Controlled Clinical Trial
Brief Title: Effect of Laser Therapy Versus Anterior Re-positioning Splint in the Treatment of Disc Displacement With Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Elzawahry, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2015-02-25
Record Dates: First submitted 2018-06-09; First posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Temporomandibular Joint Disorders
Keywords: laser therapy; anterior re-positioning splint
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Laser Therapy; Low-Level Light Therapy; Occlusal Splints

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Laser therapy (Experimental): 12 laser sessions over 3 months
  Interventions: Device: Laser therapy
- anterior re-positioning splint therapy (Active Comparator): anterior re-positioning splint worn for 8 hours during night time for 3 months
  Interventions: Device: anterior re-positioning splint
- inactive laser therapy (Placebo Comparator): placebo laser for 12 sessions over 3 months
  Interventions: Device: inactive Laser therapy

INTERVENTIONS:
Device: Laser therapy — epic model biolase with an output of 4W, 1800 J wavelength with a continuous Laser mode.
  Other Names: low-level Laser therapy; Biolase laser device
  Arms: Laser therapy
Device: anterior re-positioning splint — hard acrylic anterior re-positioning splint
  Other Names: occlusal splint; TMD splint
  Arms: anterior re-positioning splint therapy
Device: inactive Laser therapy — sham Laser, with inactive beam
  Arms: inactive laser therapy

SUMMARY:
comparing the effects of Laser therapy with anterior re-positioning splint and a placebo group on clinical signs and symptoms of temporo-mandibular dis-function and assessing articular disc morphology and configuration with magnetic resonance imaging.

DETAILED DESCRIPTION:
to compare the clinical effects of Laser therapy as assessed with research diagnostic criteria of temporo-mandibular disorders to a group that received anterior re-positioning splint therapy and a control group that received placebo Laser. Diagnosis for disc displacement with reduction was performed with magnetic resonance imaging before treatment. assessment of the clinical and MRI findings was again performed after a 3 months observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having TMD in the form of disc displacement with reduction as verified from signs and symptoms during clinical examination and confirmed from the MRI.
2. Good general health: The patient must be medically free from any systemic disease or health problems.
3. Adult patients 18 years old and above.
4. No previous orthodontic treatment.
5. No previous TMJ treatment or surgery.

Exclusion Criteria:

1. Patients with multiple missing posterior teeth.
2. Muscle pain due to systemic disease.
3. Dental related pain.
4. Congenital abnormality, neoplasia or acute trauma.
5. Previous TMJ treatment or surgery.
6. Any medical condition that prohibits MRI acquisition.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Level of temporomandibular joint pain: assessed by using subjective visual analogue scale | 3 months
  current level of temporomandibular joint pain assessed by using subjective visual analogue scale from 1 to 10 according to the research diagnostic criteria of temporomandibular disorders diagnostic sheets, zero indicates no pain, while 10 indicates the worst pain

SECONDARY OUTCOMES:
click: joint sound | 3 months
  joint sound., it is a binary measurement assessed by hand palpation
limitation of mandibular movements | 3 months
  mouth opening, measured between the incisal edges of upper and lower incisors using a digital caliper, right and left mandibular movements, measured from upper dental midline to lower dental midline using a digital caliper.
disc recapture | 3 months
  change in articular disc morphology and configuration using two dimensional measurements on a DICOM viewer software including both linear and angular measurements in relation to cartesian coordinates X and Y

CONTACTS AND LOCATIONS:
Overall Officials: Mona S Fayed, PHD, Study Director — Professor of Orthodontics, Faculty of Dentistry, Cairo Universitye

IPD SHARING:
Plan to Share IPD: Undecided